The effect of individualized analgesia on respiratory adverse events after adenotonsillectomy in Children

-randomized double-blind controlled trial

## Statistical Analysis Plan

In this study, the SPSS 23.0 (Statistical Package for Social Sciences, IBM) was used to analyze the data. The measurement data are tested by normality, and the normal distribution is expressed as the mean  $\pm$  standard deviation; if the distribution is not normal, it is represented by the median and range interquartile. The measurement data with normal distribution and homogeneity of variance uses t test, if heterogeneity of variance, use thenonparametric test; Chi square test was used to compare the count data. The data of heart rate, blood pressure and pain score were analyzed by variance analysis of repeated measurement data. Kaplan-Meier method was used to analyze the survival status of two groups patients with postoperative pain status after operation, plot the survival curve and compare the median survival time of Cheops > 6.